CLINICAL TRIAL: NCT05282355
Title: Astaxanthin Reduces Exercising Heart Rate by 7% in Overweight Individuals.
Brief Title: Astaxanthin Reduces Exercising Heart Rate.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AX2021
Record Dates: First submitted 2022-02-21; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Flexibility
Keywords: substrate oxidation; lactate; supplement
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants were blinded to either the supplement or placebo. The capsules were identical in appearance and size. Blinding was accomplished via an investigator not directly involved with data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): The astaxanthin group received 12 mg/day of astaxanthin. Each capsule contained 6 mg of astaxanthin and sunflower oil, and each subject ingested one capsule in the morning and one in the evening.
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): The placebo group ingested two capsules per day, one in the morning and one in the evening. Each capsule contained sunflower oil and mimicked the size and appearance of the astaxanthin supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin — Our aim was to examine the impact astaxanthin would have, if any, on markers of metabolic flexibility in overweight individuals in comparison to a placebo.
  Arms: Astaxanthin
Dietary Supplement: Placebo — To have adequately test the effects of astaxanthin, we provided one group a placebo matched in appearance and taste.
  Arms: Placebo

SUMMARY:
Briefly, this study involved 2 trials: baseline (Trial 1) and post-astaxanthin intervention (Trial 2). Both trials included participants completing a graded exercise test while connected to a metabolic cart, to measure cardiorespiratory measures. Between trials, participants were supplemented with either 12 mg of astaxanthin or placebo for 4 weeks. It was hypothesized astaxanthin supplementation would increase rates of fat oxidation, while decreasing carbohydrate oxidation and blood lactate accumulation.

DETAILED DESCRIPTION:
METHODS

Experimental Design

The current study implemented a double-blind, between-subject study design with dependent variables examined at multiple timepoints across each trial. To best observe changes in our selected dependent variables, subjects reported to the laboratory on two separate occasions (i.e. pre-post) following 4 weeks of astaxanthin supplementation.

Subject Approval from the Institutional Review Board was granted before recruiting subjects (University of North Alabama, Institutional Review Board #: 20-21-071). Each subject completed a Physical Activity Readiness Questionnaire, a medical questionnaire, and provided their written and verbal consent to voluntarily participate in the present study. Inclusion criteria for each subject included the following: 1) between the ages of 18-45; 2) free of any cardiometabolic disease medication; 3) classified as overweight with a bodyfat percent of ≥ 20% for males and ≥ 25% for females; 4) and not currently pregnant or actively trying to become pregnant. Additionally, subjects eliminated all dietary supplements at least two weeks prior to the start of the study. Using G-Power software and changes to bodyfat as a primary dependent variable, we determined a priori that 20 subjects would be sufficient to achieve a desired power of 0.85, using a moderate-high effect size, and an alpha level set at 0.05. Although 46 individuals were recruited, only 21 fit the inclusion criteria and were randomized into either an astaxanthin or placebo group following their first visit. Due to two participants withdrawing from the study as a result of health concerns not related to the study procedures, 19 subjects were included in statistical analysis.

Preliminary Data During the first visit, subjects had their body composition assessed via bioelectrical impedance analysis as well as height, mass, and blood pressure by the same, trained investigator pre-post intervention. Following the collection of anthropometric data, subjects who met inclusion and exclusion criteria were then asked to attempt to maintain their current dietary habits for the duration of the intervention. Dietary intake was then recorded pre-post intervention via 3-day food logs which consisted of 2 weekdays and 1 weekend day (i.e. Thursday, Friday, Saturday) to better reflect typical intakes. Subjects met with the primary investigator and were instructed how to complete the food logs, regarding quantity size and liquid amount estimations. Total energy intake, carbohydrate, protein, and fats were analyzed for nutrient amounts using MyFitnessPal and were then used in statistical analysis.

Experimental Trials (Trials 1-2) Following the collection of preliminary data, subjects completed a graded exercise test on a cycle ergometer. Prior to the start of exercise, subjects donned a heart rate monitor, established seat height, and were then connected to a metabolic cart to record cardiorespiratory measures for the calculation of fat and carbohydrate oxidation rates. Following connection to the metabolic cart, subjects sat quietly for 5 min to collect resting oxidation rates ('rest'). Subjects then straddled the cycle ergometer and began pedaling at an initial 30 W (females) or 50 W (males) for 5 min (Stage 1). For each subsequent stage, resistance increased by 15 W and lasted for 5 min (Stages 2-5). Following completion of 5 stages (90 W total for females and 110 W total for males), resistance then increased by 15 W every minute, until volitional exhaustion was achieved and the subjects' volume of oxygen (VO2) peak was recorded. The present protocol was pilot tested (n = 6) prior to the initiation of the present study and determined by the investigative team as acceptable for non-exercising and overweight individuals to all complete with minimal fluctuation in heart rate (±2 bpm) during the last min of each stage.

During the last 30 s of each stage, subjects had their finger pricked (detailed further below) for the measurement of capillary lactate and glucose. Furthermore, heart rate and overall ratings of perceived exertion were recorded at the end of each stage. Due to the collection of oxidation rates, subjects were required to fast for 5 h and avoid alcohol consumption for 48 h prior to each trial. Subjects were also required to abstain from caffeine on the day of testing and avoid strenuous lower body exercise 48 h prior to each experimental trial.

Fat and Carbohydrate Oxidation Rate Measurements All cardiorespiratory measures were averaged from expired gas collected by the metabolic cart. The first 240 seconds of each stage were excluded and the remaining 60 seconds were recorded using breath-by-breath data and averaged in two, 30-second cycles. Stoichiometric equations were utilized when measuring total fat and carbohydrate oxidation rates (g · min-1). These equations assumed protein oxidation rates were negligible (~5%) and therefore, were ignored.

Fat oxidation (g ∙ min-1) = 1.67 VO2 (L ∙ min-1) - 1.67 VCO2 (L ∙ min-1) Carbohydrate oxidation (g ∙ min-1) = 4.55 VO2 (L ∙ min-1) - 3.21 VCO2 (L ∙ min-1)

Lactate and Glucose Concentration Measurement At the end of each stage during the graded exercise test, a sample of capillary blood was collected from the subjects' finger. The subjects had their finger wiped with an alcohol swab and then allowed to air dry prior to a prick with a self-withdrawing safety lancet. The first drop of blood was wiped away and the second drop of blood was analyzed using a Lactate Plus Meter Blood Analyzer. Additionally, capillary blood glucose concentrations were analyzed using a Precision Xtra Blood Glucose Analyzer

. Supplementation Schedule The supplementation intervention was scheduled following Trial 1 and took place for 4 weeks before subjects reported back to the laboratory for Trial 2. Subjects were randomly assigned to supplement with either 12 mg of encapsulated astaxanthin (astaxanthin and sunflower oil; 6 mg per capsule) or placebo (sunflower oil only) daily in the form of two gel capsules. Subjects were advised to ingest one capsule in the morning and one capsule at night. Both the astaxanthin and placebo pills were similar in appearance (red and oval shaped) and size and all supplements were provided by AstaReal.

ELIGIBILITY:
Inclusion Criteria:

* Free of any cardiometabolic disease medication
* Classified as overweight - body fat % ≥ 20% (M) and ≥ 25% (F)
* Exclude dietary supplements for 2 weeks prior to start of study

Exclusion Criteria:

* If there is a chance of pregnancy
* body fat % < 20% (M) and < 25% (F)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Changes to substrate oxidation rates | Up to 4 weeks
  Substrate oxidation rates reflect cellular utilization of carbohydrates and lipids at rest and during exercise. If changes exist from astaxanthin supplementation, they would manifest themselves likely via increases to rates of fat oxidation at all stages and a subsequent decrease in carbohydrate oxidation rates at each stage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Alabama, Department of Kinesiology, Florence, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Unless required, we do not plan on sharing our subjects data, even though the data is coded. Since this study is being registered post-completion, we did not make our subjects aware their data may be shared outside of our research team and therefore, we find this a potential conflict of ethical consideration for our subjects.